CLINICAL TRIAL: NCT05869019
Title: Developing and Implementing the Self-Efficacy Scale of Mothers of Premature Infants Based on Individualized Developmental Care
Brief Title: Self-efficacy Scale for Mothers of Premature Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayşegül Karaca, nurse, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOKTORA TEZ AYSEGUL
Record Dates: First submitted 2023-04-10; First posted 2023-05-22 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Baby Care
Keywords: prematüre; mother; scale
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- providing education (Experimental): There are two groups, training and non-training.
  Interventions: Other: education

INTERVENTIONS:
Other: education — Premature baby care training will be provided.

SUMMARY:
The aim of this study is to develop a scale to determine the self-efficacy of mothers of premature infants in individualized developmental care practices.

This study consists of two stages. In the first stage, it is planned to develop a scale to determine the self-efficacy levels of mothers of premature babies based on individualized developmental care. In the second stage, the scale will be applied. At this stage, families will be trained for individualized developmental care and the effectiveness of the education will be evaluated through the developed scale.

For the first stage of the study, it is stated in the literature that at least 5 times the number of items should be taken in determining the sample size during the scale development stage, and 10 times in order to increase the reliability of the scale. In this study, after creating the scale items, a pilot application will be made with 3 mothers. Feedback will be received from mothers regarding the clarity of the questions and the scale will be finalized according to the feedback received. Then, the scale will be applied to the participant with a size of at least 10 times the number of scale items.

For the second phase of the study, firstly, a preliminary application will be made with 10 mothers who meet the inclusion criteria and agree to participate in the study. The number of samples to be taken for the second stage of the research will be determined by performing power analysis with the findings obtained. Mothers included in the preliminary application will not be included in the study. It is planned to use stratified block randomization method in the study. First, mothers will be stratified according to their education level and the total number of children they have, then an equal number of (blocking) mothers will be assigned to each group.

Data will be collected after obtaining written permission from the institution where the research will be conducted. "Descriptive Information Form", "Informed Voluntary Consent Form" prepared by the researchers and "Individualized Developmental Care Based Premature Baby Mothers' Self-Efficacy Scale" will be used in data collection.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of premature babies whose babies were discharged from the Neonatal Intensive Care Unit (NICU) (training will be given immediately after the baby is discharged),
* Continuing prematurity of the baby according to the corrected age,
* Full-time care of the baby at home by the mother,
* Mothers can speak and understand Turkish,
* Voluntary written and verbal informed consent was obtained from the mothers.

Exclusion Criteria:

* Being a term baby
* The mother has an ongoing psychological diagnosis,
* The mothers' unwillingness to continue working at any stage of the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study will be conducted with mothers of premature babies.
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Infant care activities of mothers of premature infants will be evaluated with the Self-Efficacy Scale for Mothers of Premature Infants Based on Individualized Developmental Care. | On the first day of the babies' discharge, face-to-face interviews will be provided with mothers.
  Implementing the Self-Efficacy Scale of Mothers of Premature Infants Based on Individualized Developmental Care

SECONDARY OUTCOMES:
Infant care activities of mothers of premature infants will be evaluated with the Self-Efficacy Scale for Mothers of Premature Infants Based on Individualized Developmental Care. | Face-to-face interviews will be provided with mothers 15 days after their babies are discharged from the premature intensive care unit.
  Implementing the Self-Efficacy Scale of Mothers of Premature Infants Based on Individualized Developmental Care

IPD SHARING:
Plan to Share IPD: No